CLINICAL TRIAL: NCT06711393
Title: The Effectiveness of Exergaming (YetiHome®) Versus Traditional Exercise for Older People Mobility and Balance: Protocol of the Randomized Intervention Trial
Brief Title: The Effectiveness of Exergaming for Older People Mobility and Balance
Acronym: YetiExergame
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Sari Arolaakso, Senior Lecturer, PhD student, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 61/2023
Record Dates: First submitted 2024-11-25; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Mobility Limitation
Keywords: Older adults; Balance; Mobility limitation; Preclinical mobility limitation
MeSH Terms: conditions — Mobility Limitation | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exergaming group (Experimental): Exergaiming group plaing games during intervention period
  Interventions: Other: Exercise
- Control group (Active Comparator): Regular exercise without exergaming
  Interventions: Other: Exercise as usual

INTERVENTIONS:
Other: Exercise — Traditional home exercise including balance and muscle strength training 15 minutes at the time and three times over the week. In addition, game-based exercises 15 minutes at the time and three times over the week.
  Arms: Exergaming group
Other: Exercise as usual — Traditional home exercise including balance and muscle strength training 15 minutes at the time and three times over the week without exergaming.
  Arms: Control group

SUMMARY:
The mobility problems of older people are often related to the decrease of functional capacity and health [1], weakened physical condition, attitude to life and fear of falling [2]. Relatively little research has been done on the possibilities and effectiveness of exergaming on the mobility of old people. Interventions that include exergaming have been found to motivate and increase commitment to rehabilitation [3], to improve mobility, balance [4], performance in daily activities and independence [5].

The aim of randomized intervention trial is to find out the effect of physical exercises performed on the technological device (YetiHome®) on identified preclinical movement problems during a 2-month follow-up period. The goal is to produce information about the effectiveness of gamified physical exercises in preventing movement problems and supporting older people living at home.

This study investigates the effectiveness of the YetiHome in improving the physical functioning of older people. YetiHome is an assistive technology device developed for special groups. YetiHome is a small interactive touchscreen tablet with 27" screen and with Android operating system and it includes numerous applications. Added exergaming solution for the balance training. There is no previous scientific research on the effectiveness of the YetiHome on the mobility problems and activity of the community-dwelling older people living independently at home.

The aim of randomized intervention trial is to find out the effect of physical exercises performed on the technological device (YetiHome®) on identified preclinical movement problems during a 2-month follow-up period. The goal is to produce information about the effectiveness of gamified physical exercises in preventing movement problems and supporting older people living at home.

This study investigates the effectiveness of the YetiHome in improving the physical functioning of older people. YetiHome is an assistive technology device developed for special groups. YetiHome is a small interactive touchscreen tablet with 27" screen and with Android operating system and it includes numerous applications. Added exergaming solution for the balance training. There is no previous scientific research on the effectiveness of the YetiHome on the mobility problems and activity of the community-dwelling older people living independently at home.

DETAILED DESCRIPTION:
Sample size calculation was completed based on an effect size of 0.35 (power = 0.80; α= 0.05). Assuming a 35% attrition rate, a total of 100 participants will be recruited (50 people in a control group and 50 people in the intervention group). The target group is 75 old people, who are not covered by social and health services and who have received a preventive home visit in the region of Kemi in northern Finland. The intervention groups consist of people who have been found to have preclinical mobility problems during a preventive home visit.

After being informed about the study all suitable participants of the preventive home visit willing to participate in this study will undergo baseline functional testing on week 0. Same functional measurements will be conducted after two-month intervention period. Baseline data collection of functional capacity utilizes the structured questionnaire (HEKO-tool), whose functional assessment targets are bridged to the ICF classification (International Classification of Functioning, Disability and Health). Data is collected on everyday activities as well as mental-wellbeing, social-wellbeing and risk of falls. In the second phase, the physical performance was assessed by a One-Leg Balance test (OLB) and Short Physical Performance test (SPPB) combined with a mobile solution developed to measure balance, AinoneBalance. The AinoneBalance application utilizes Romberg's standardized test. The participants were randomized into a game group and a control group. The gaming group received a YetiHome® device at home and instructions for the traditional exercise. The control group only received instructions for the traditional exercise.

ELIGIBILITY:
Inclusion Criteria:

* Living at home.
* Not a user of health and social services.
* Sufficient cognitive ability to do exercises independently.

Exclusion Criteria:

* Risk of hip fracture and inability to perform exercise independently.

Ages: 75 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-27 (Estimated); Primary Completion 2024-12-20 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Balance Short Physical Performance Battery (SPPB) | From baseline to the end of intervention at 8 weeks
  Short Physical Performance Battery (SPPB), Scores range from 0 to 12. The lower the SPPB total score, the greater the risk of future mobility.
One Leg Balance (OLB) | From baseline to the end of intervention at 8 weeks
  AinoneBalance -solution, Movement path length. Standing 10 seconds with feet together, semi tandem, tandem, the eyes open and closed, on hard and soft surface.
Mobility | From enrollment to the end of treatment at 8 weeks
  Short Physical Performance Battery (SPPB), Scores range from 0 to 12. The lower the SPPB total score, the greater the risk of future mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Satu Elo Elo, PhD, Adjunct professor, Principal lecturer, Study Director — University of Oulu
Locations (1):
- Research unit of health sciences and technology, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neumann S, Meidert U, Barbera-Guillem R, Poveda-Puente R, Becker H. Effects of an Exergame Software for Older Adults on Fitness, Activities of Daily Living Performance, and Quality of Life. Games Health J. 2018 Oct;7(5):341-346. doi: 10.1089/g4h.2017.0079. PMID 30325234
- [Background] Pacheco TBF, de Medeiros CSP, de Oliveira VHB, Vieira ER, de Cavalcanti FAC. Effectiveness of exergames for improving mobility and balance in older adults: a systematic review and meta-analysis. Syst Rev. 2020 Jul 18;9(1):163. doi: 10.1186/s13643-020-01421-7. PMID 32682439
- [Background] Oesch P, Kool J, Fernandez-Luque L, Brox E, Evertsen G, Civit A, Hilfiker R, Bachmann S. Exergames versus self-regulated exercises with instruction leaflets to improve adherence during geriatric rehabilitation: a randomized controlled trial. BMC Geriatr. 2017 Mar 23;17(1):77. doi: 10.1186/s12877-017-0467-7. PMID 28330455
- [Background] Pauelsen M, Nyberg L, Roijezon U, Vikman I. Both psychological factors and physical performance are associated with fall-related concerns. Aging Clin Exp Res. 2018 Sep;30(9):1079-1085. doi: 10.1007/s40520-017-0882-9. Epub 2017 Dec 20. PMID 29264814
- See also: GeroNursing Center, Research unit of health sciences and technology, University of Oulu — https://geronursing.fi/in-english/